CLINICAL TRIAL: NCT04519255
Title: Single-center, Open, Prospective, Randomized Pilot Study for Quantitative Analysis of Whole Body Inflammatory Lesions in Recovered COVID-19 Patients by 18F-FDG-PET/CT
Brief Title: Study for Quantitative Analysis of the Recovered COVID-19 Patients by 18F-FDG-PET/CT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FZYX.008
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-07

CONDITIONS: PET/CT; COVID-19; Respiratory Function; Inflammatory Lesions
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Screening of clinically cured patients with severe COVID-19: ①Patients with severe COVID-19 cure were determined based on nucleic acid tests, CT examinations, and clinical criteria; ②Age > 18 years, age < 85 years, no gender restriction; ③ All had received COVID-19 drug therapy; ④ ECOG of general condition score: 0-2; No dysfunction of main viscera; Oxygen partial pressure ≥10.64kPa; White blood cells ≥4×109/L; Blood routine hemoglobin ≥9.5g/dL; The absolute count of neutrophils ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; Creatinine ≤1.25 times the upper limit of normal value; The creatinine clearance rate was ≥60ml/min; ⑤ Can obtain complete follow-up information, understand the situation of this study and sign informed consent.
- Screening of clinically cured patients with mild COVID-19: ①Patients with mild COVID-19 cure were determined based on nucleic acid tests, CT examinations, and clinical criteria; ②Age > 18 years, age < 85 years, no gender restriction; ③ All had received COVID-19 drug therapy; ④ ECOG of general condition score: 0-2; No dysfunction of main viscera; Oxygen partial pressure ≥10.64kPa; White blood cells ≥4×109/L; Blood routine hemoglobin ≥9.5g/dL; The absolute count of neutrophils ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; Creatinine ≤1.25 times the upper limit of normal value; The creatinine clearance rate was ≥60ml/min; ⑤ Can obtain complete follow-up information, understand the situation of this study and sign informed consent.
- Healthy people who are not infected with COVID-19: ① Volunteers who are not infected with COVID-19; ②Age > 18 years, age < 85 years, no gender restriction; ③ ECOG of general condition score: 0-2; No dysfunction of main viscera; Oxygen partial pressure ≥10.64kPa; White blood cells ≥4×109/L; Blood routine hemoglobin ≥9.5g/dL; The absolute count of neutrophils ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; Creatinine ≤1.25 times the upper limit of normal value; The creatinine clearance rate was ≥60ml/min; ④ Can obtain complete follow-up information, understand the situation of this study and sign informed consent.

SUMMARY:
In this study, clinically cured patients with severe COVID-19 were used to evaluate the therapeutic effect of COVID-19 and the recovery and health status of patients over time with highly sensitive PET/CT imaging technology. At the same time, PET/CT whole body scan, dynamic imaging and mathematical dynamic model were combined to evaluate the functions of the heart, lung, liver, kidney, brain and other important organs and the outcome of inflammatory lesions in clinically cured COVID-19 patients.

DETAILED DESCRIPTION:
Covid-19 (Corona Virus Disease 2019, COVID-19), referred to as "COVID-19", refers to the pneumonia caused by novel Coronavirus 2019 (2019-NCOV/SARS-COV-2) infection. The clinical manifestations of the new patients were fever, fatigue and dry cough, while the symptoms of upper respiratory tract such as nasal congestion and runny nose were rare. Hypoxia occurs. About half of the patients developed dyspnea after one week, and in severe cases, the rapid progression was acute respiratory distress syndrome, septic shock, metabolic acidosis that was difficult to correct, and coagulation dysfunction. After the outbreak of COVID-19 in China, the National Health Commission issued the Diagnosis and Treatment Plan for COVID-19. By analyzing the epidemic situation and research progress, it organized experts to timely revise the diagnosis and treatment plan based on the analysis, study and summary of the previous medical treatment work.The discharge criteria for COVID-19 patients notified by the National Health Commission are remission of clinical symptoms, normal body temperature, normal CT, and negative nucleic acid tests for both tests. So far, the COVID-19 epidemic in China has been well under control. According to the latest statistics, 84,311 cases have been confirmed in total, and 1,433 cases have been confirmed so far.But studies (the latest from Dena Goffman's team, published in the NEJM) suggest that as many as 88 percent of coVID-19 patients are asymptomatic. Do cured patients leave the hospital with a percentage of asymptomatic patients?In addition, covid-19 cured patients in some regions turned positive again after discharge, indicating that long-term follow-up monitoring is of great significance for cured and discharged patients in addition to routine isolation observation!Moreover the literature at home and abroad other viral infections (such as hepatitis b, HIV, etc.) to cure patients found that the virus may lurk for a long time, the virus quantity contained in a very low level, the conventional detection method is difficult to detect, at the appropriate incentives can lead to attack, so for the new crown cure patients need close monitoring of systemic inflammation related lesions, and the situation of the latent virus.However, we still face many problems and challenges. For example, according to the latest data published by Dena Goffman's team in NEJM, the proportion of asymptomatic patients is as high as 88%, so the screening of asymptomatic patients is crucial.In many places, COVID-19 patients cured turn positive again after discharge. Therefore, it is of great significance to explore the mechanism of COVID-19 turning negative after discharge and evaluate the effect of novel Coronavirus and COVID-19 on patients' later recovery. Explore and develop more efficient and sensitive clinical detection methods to evaluate the treatment effect of covid-19 patients.

Positron emission computed tomography imaging technique is a nuclear medicine clinical diagnosis of advanced imaging techniques, can be shown on the in vivo biological molecules (such as 18 F- FDG, tracer nuclide labeled glucose molecules) metabolism, receptors and neurotransmitter activity of new functional imaging techniques, has been widely used in many kinds of disease diagnosis and differential diagnosis, a judgment, curative effect evaluation, viscera function research and development of new drugs, etc. Compared with traditional anatomical structure imaging, functional imaging PET has the following advantages: (1) High sensitivity. According to the test, PET molecular probe can pick up molecular events at the level of PM-NM in vivo. (2) High specificity, for the PET selected molecular probe, can only imaging the target molecules, for the same family of receptors, because the binding degree difference can be specifically distinguished; (3) Whole-body imaging, that is, one time PET imaging can obtain images of all regions of the whole body, and through the analysis can obtain the dynamic information of the metabolic changes of human tissues over time, which is of great significance for the research, prevention and evaluation of diseases.In particular, PET/CT scan provides a more reliable means of systemic monitoring for viruses that are lurking in all hidden parts of the body. (4) Security is good, although there are some radioactive nuclide PET need, but the amount of nuclide rarely used with short half-life, through two aspects of physical decay and biological metabolism function, in a very short time, client retention, a PET general inspection of radiation dose is far less than the conventional CT examination of a part, and safe and reliable.

ELIGIBILITY:
Inclusion Criteria:

Screening of clinically cured patients with severe COVID-19:

* Patients with severe COVID-19 cure were determined based on nucleic acid tests, CT examinations, and clinical criteria;
* Age > 18 years, age < 85 years, no gender restriction;
* All had received COVID-19 drug therapy;
* ECOG of general condition score: 0-2; No dysfunction of main viscera; Oxygen partial pressure ≥10.64kPa; White blood cells ≥4×109/L; Blood routine hemoglobin ≥9.5g/dL; The absolute count of neutrophils ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; Creatinine ≤1.25 times the upper limit of normal value; The creatinine clearance rate was ≥60ml/min;
* Can obtain complete follow-up information, understand the situation of this study and sign informed consent.

Screening of clinically cured patients with mild COVID-19:

* Patients with mild COVID-19 cure were determined based on nucleic acid tests, CT examinations, and clinical criteria;
* Age > 18 years, age < 85 years, no gender restriction;
* All had received COVID-19 drug therapy;
* ECOG of general condition score: 0-2; No dysfunction of main viscera; Oxygen partial pressure ≥10.64kPa; White blood cells ≥4×109/L; Blood routine hemoglobin ≥9.5g/dL; The absolute count of neutrophils ≥1.5×109/L; Platelet count ≥100×109/L; Total bilirubin ≤1.5 times the upper limit of normal value; Creatinine ≤1.25 times the upper limit of normal value; The creatinine clearance rate was ≥60ml/min;
* Can obtain complete follow-up information, understand the situation of this study and sign informed consent.

Exclusion Criteria:

* Poorly controlled diabetics (fasting glucose level and GT;200 mg/dL);
* Any other malignancy within 5 years;
* Breastfeeding and/or pregnant women;
* Those who are prone to severe bleeding;
* Recent severe hemoptysis, severe cough, dyspnea or patients cannot cooperate;
* Severe emphysema, pulmonary congestion and pulmonary heart disease;
* The researchers believe that the subjects may not be able to complete the study or comply with the requirements of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 cured were determined based on nucleic acid tests, CT examinations, and clinical criteria. The age of patient were between 18 and 85 years, meanwhile in Zhuhai they were confirmed as COVID-19, cured and all received by COVID-19 drug therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of clinically cured patients with severe COVID-19 | 6 months
  Count the number of clinically cured patients with severe COVID-19
Number of clinically cured patients with mild COVID-19 | 6 months
  Count the number of clinically cured patients with mild COVID-19
Number of healthy people who are not infected with COVID-19 | 6 months
  Count the number of healthy people who are not infected with COVID-19
Ki comparison between the severe, the mild and the healthy | 12 months
  Ki of the severe, the mild and the healthy were calculated and compared
SUVmax comparison between the severe, the mild and the healthy | 12 months
  SUVmax of the severe, the mild and the healthy were calculated and compared

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shan, Ph.D, Study Chair — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Hongjun Jin, Zhuhai, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao J, Liu J, Bi L, Huang Y, Wang L, Zhang F, Wang Y, Jin H. The imaging quantification of multiple organs by dynamic 18F-FDG PET/CT in discharged COVID-19 patients: A prospective pilot study. Int J Med Sci. 2022 Sep 6;19(10):1539-1547. doi: 10.7150/ijms.73801. eCollection 2022. PMID 36185330